CLINICAL TRIAL: NCT06467708
Title: Delivering Transcutaneous Auricular Neurostimulation (tAN) to ICU Patients With Traumatic Brain Injury (tAN-TBI)
Brief Title: Transcutaneous Auricular Neurostimulation for ICU Patients With Traumatic Brain Injury
Acronym: tAN-TBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Alex Valadka, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0360
Record Dates: First submitted 2024-05-29; First posted 2024-06-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-01

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Transcutaneous auricular neurostimulation (tAN)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: TBI patients in the ICU with Glasgow Coma Scale score of 12 or below and acute traumatic intradural blood on head CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Determine the effect of tAN on serum concentrations of inflammatory mediators in TBI patients (Experimental): Subjects will receive treatment upon providing informed consent and will undergo transcutaneous auricular neurostimulation (tAN) once daily during their ICU stay, with the treatment duration not exceeding 10 days. Two blood samples will be collected daily: one before the tAN session and another two hours after the session. Participant data will be collected daily throughout the ICU stay. Additionally, surveys will be collected from registered nurses providing direct care to TBI patients enrolled in the tAN-TBI study to assess the compatibility of tAN with patient care processes in the ICU.
  Interventions: Device: Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN)

INTERVENTIONS:
Device: Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) — This method of simultaneous vagal and trigeminal stimulation via the external ear is known as transcutaneous auricular neurostimulation (tAN), as the targets of electrical stimulation include the auricular branch of the vagus nerve (ABVN) and auriculotemporal nerve (ATN), which is a branch of the mandibular division of the trigeminal nerve. Electrodes applied to select dermatome regions can target ear neural structures and deliver non-invasive vagus nerve stimulation (VNS) and trigeminal nerve stimulation (TNS).

SUMMARY:
The overarching goal of this pilot study is to assess the feasibility and safety of transcutaneous auricular neurostimulation (tan) in ICU patients with TBi and to determine the effect of tan on serum markers of inflammation. exploratory analyses will examine effects on such physiological parameters as blood pressure, heart rate, and intracranial pressure (iCP), as well as measures of neurological function.

DETAILED DESCRIPTION:
This is a single-center, open-label, nonrandomized investigation. TBI patients with a post resuscitation Glasgow Coma Scale (GCS) score of 12 or less (commonly described as moderate or severe TBI) and acute traumatic intradural blood on head CT scan will be screened upon admission to the ICU at Parkland Memorial Hospital. It is expected that all or almost all subjects will be in the Neuroscience or Surgical ICU. Consent for participation will be sought from the subject's legally authorized representative. Exception from informed consent or waiver of consent will not be part of this study.

tAN will begin as soon as feasible after subject enrollment. Immediately prior to this intervention, vital signs, neurologic status, and other clinical parameters will be recorded, and pre-tAN blood will be collected for measurement of serum inflammatory markers. tAN will be administered for 30 minutes under the supervision of a member of the research team. After 30 minutes (just prior to stopping tAN), the same clinical parameters that were recorded at baseline will again be recorded then tAN will be stopped. Approximately two hours after tAN has ended, a post-tAN blood sample will be collected for measurement of the same inflammatory markers as in the pre-tAN blood sample. At each timepoint for blood collection, additional blood may be collected for banking and future analyses.

Patients will undergo research blood draws and tAN stimulation for a maximum of 10 days. Research-related procedures will not exceed this 10-day period.

ELIGIBILITY:
Inclusion Criteria:

1. Post-resuscitation GCS score 12 or below and acute trauma-related intradural blood on head CT scan after TB
2. Age 18 years or older (pediatric trauma patients are not routinely transported to Parkland)
3. Consent from legally authorized representative

Exclusion Criteria:

1. Hemodynamic instability
2. Expected imminent mortality because of overwhelming neurological and/or systemic injury
3. Unclear neurological status because of paralytic medications or intoxication with ethanol or other drugs
4. Presence of other electrical stimulation devices (pacemaker, cochlear prosthesis, neurostimulator, etc.)
5. Abnormal ear anatomy or ear infection
6. Participant is pregnant or lactating
7. Any other significant medical or psychosocial problems that, in the opinion of the investigator, would potentially cause harm to the participant, impact their ability to participate, or influence the results of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-02-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Survey nursing attitudes towards daily tAN and the compatibility of tAN with standard patient care activities in the ICU; Examine the safety of tAN in ICU patients. | Registered nurses can complete the Sparrow Ascent ICU User Acceptance Questionnaire at Day 1- Day 10, or before the TBI patient is discharged from the hospital, or ICU. It may not be completed on Day 11 or after the patient has been discharged.
  Registered nurses providing direct care to ICU patients receiving tAN will be asked to complete the Sparrow Ascent ICU User Acceptance Questionnaire to assess the compatibility of tAN with patient care.
Determine the effect of tAN on serum concentrations of inflammatory mediators in TBI patients. | TBI patients will receive tAN stimulation once per day and will not exceed 10 days.
  Every effort will be made to initiate tAN as soon after injury as possible in order to capture early postinjury data on the effectiveness of tAN and to inform the design of future studies.
Explore the effect of tAN on Blood Pressure | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Blood pressure (mmHg) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Heart Rate | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Heart rate (bpm) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Respiratory Rate (and ventilator settings and use of noninvasive oxygenation and ventilation if applicable) | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Respiratory rate (bpm) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Temperature | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Temperature (°C/°F) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Intracranial pressure | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Intracranial pressure (mmHg) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Brain Tissue Oxygen Tension (PbtO2) | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Brain Tissue Oxygen Tension (mmHg) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Glasgow Coma Scale (GCS) (and any sedatives or analgesics that could affect neurological assessment) | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  GCS (and any sedatives or analgesics that could affect neurological assessment) will be checked twice daily, pre-tAN and 30 minutes post-tAN. Scale from 3 to 15, where 3 represents deep unconsciousness and 15 indicates full consciousness.
Explore the effect of tAN on Pupillary Diameter | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Pupillary Diameter (mm) will be checked twice daily, pre-tAN and 30 minutes post-tAN
Explore the effect of tAN on Neurological Pupil index (NPi) via pupillometry | Data will be collected upon consent, twice daily from Day 1 to Day 10, or until the patient is discharged from the hospital. Data will not be collected past 10 days.
  Neurological Pupil index (NPi) via pupillometry dimensionless index, typically ranging from 0 to 5. This will be checked twice daily, pre-tAN and 30 minutes post-tAN

CONTACTS AND LOCATIONS:
Overall Officials: Alex Valadka, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States